CLINICAL TRIAL: NCT04089540
Title: New Intubation Method to Achieve Circulatory Stability and to Reduce Number of Intubation Attempts in Neonates. A Pilot Study
Brief Title: New Intubation Method to Achieve Circulatory Stability and to Reduce Number of Intubation Attempts in Neonates
Acronym: NOONA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NOONA
Record Dates: First submitted 2019-09-05; First posted 2019-09-13 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Intubation; Difficult or Failed; Preterm Infant; Term Infant
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group: New intubation method (Experimental): In the new intubation method the respirator is connected to the tube prior to insertion into the mouth (oral intubation) or into the nose (nasopharyngeal intubation). Therefore an oxygen flow is already administered via the tube during the intubation process.
  Interventions: Procedure: New intubation method
- Control group: Conventional intubation (Other): In the control group the respirator is connected to the tube and ventilation is started after the insertion of the tube into the trachea. Therefore there is no oxygen flow administered during the intubation process.
  Interventions: Procedure: Conventional intubation method

INTERVENTIONS:
Procedure: New intubation method
  Arms: Study group: New intubation method
Procedure: Conventional intubation method
  Arms: Control group: Conventional intubation

SUMMARY:
This is a randomized controlled pilot study investigating a new intubation method in newborn infants. In contrast to the conventional intubation method, in the new method the respirator is connected to the tube prior to insertion into the mouth (oral intubation) or into the nose (nasopharyngeal intubation). As a result, an oxygen flow is already administered via the tube during the intubation process. Heart rate, arterial oxygen saturation (SpO2) and cerebral tissue oxygenation (using near-infrared spectroscopy) are recorded in both the study and control groups during intubation.

Hypothesis

* The new intubation method is safe
* The new intubation method leads to a reduction in the number of intubation attempts
* The new intubation method leads to a reduction of desaturations and bradycardia during intubation
* In the long term, it could lead to a reduction in morbidity and mortality

ELIGIBILITY:
Inclusion Criteria:

* Preterm and term born neonates who are hospitalized at neonatal intensive care unit, Medical University of Graz, Austria.
* Fulfillment of indication for intubation

Exclusion Criteria:

- Malformation of the upper respiratory tract

Ages: 1 Minute to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2021-01 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Number of intubation attempts | During intubation process
  Changes in the number of intubation attempts

SECONDARY OUTCOMES:
Duration of intubation process in minutes | During intubation process
  Changes in duration
Number of desaturations | During intubation process
  The number of desaturations below 80% SpO2
  The number of bradycardia below 100 beats per minute (bpm), as well as the total amount of time a patient spends less than 100 bpm.
Total amount of time of desaturations | During intubation process
  The total amount of time in seconds a patient spends below 80% SpO2.
  The number of bradycardia below 100 beats per minute (bpm), as well as the total amount of time a patient spends less than 100 bpm.
Cerebral tissue oxygenation | 5 minutes before intubation start till 10 minutes after successful intubation
  Using near-infrared spectroscopy to monitor changes of the cerebral tissue oxygenation
Morbidity | up to 2 years
  Changes in morbidity
Mortality | up to 2 years
  Changes in mortality

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Morris, MD, Principal Investigator — Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Austria
Locations (1):
- Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Graz, Austria